CLINICAL TRIAL: NCT07394868
Title: Comparison of the Analgesic Efficacy of Combined Superficial and Deep Serratus Anterior Plane Block Versus Superficial Serratus Anterior Plane Block Following Modified Radical Mastectomy Surgery
Brief Title: Comparison of the Combined Serratus Anterior Plane Block Versus Superficial Serratus Anterior Plane Block
Status: Not yet recruiting | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Yusuf Özgüner, Principal Investigator, Ankara Etlik City Hospital
Other Study IDs: Etlik Kübra Tez
Record Dates: First submitted 2026-01-31; First posted 2026-02-06 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Pain
Keywords: Breast surgery; Multimodal analgesia; Serratus anterior plane block
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Combined superficial and deep serratus anterior plane block: Patients who will undergo combined serratus anterior plane block will be included in this group.
  Interventions: Other: Combined serratus plan block
- Superficial serratus anterior plane block: Patients who will undergo a superficial anterior plane serratus block will be included in this group.
  Interventions: Other: Superficial serratus plane block

INTERVENTIONS:
Other: Combined serratus plan block — Combined serratus plan block
  Groups: Combined superficial and deep serratus anterior plane block
Other: Superficial serratus plane block — Superficial serratus plane block
  Groups: Superficial serratus anterior plane block

SUMMARY:
Breast cancer is the most common malignancy in women; surgery is a cornerstone of breast cancer treatment, and modified radical mastectomy is one of the standard treatments. Postoperative pain can significantly reduce the quality of life in patients, and acute pain can even trigger chronic pain syndrome. Thoracic paravertebral, thoracic epidural, intercostal nerve, and interscalene brachial plexus blocks have been used for anesthesia and abiration during modified radical mastectomy, but their application is limited due to the complex nature of the procedures and serious complications. In recent years, there has been increasing interest in the newer, less invasive superficial serratus block and combined serratus block. Serratus anterior plane block (SAPB) can be applied in two ways. Deep SPB (DSPB) is applied under the serratus anterior muscle, while superficial SPB (YSPB) is applied above the serratus anterior muscle. In recent years, deep + superficial SPB, or combined SPB (KSPB), has begun to be applied in order to increase the area of effect of local anesthetics and to prevent block failure. This study aims to compare superficial and combined serratus anterior plane blocks.

DETAILED DESCRIPTION:
Breast cancer is the most common malignancy in women; surgery is a cornerstone of breast cancer treatment, and modified radical mastectomy is one of the standard treatments. Postoperative pain can significantly reduce the quality of life in patients, and acute pain can even trigger chronic pain syndrome. Thoracic paravertebral, thoracic epidural, intercostal nerve, and interscalene brachial plexus blocks have been used for anesthesia and abiration during modified radical mastectomy, but their application is limited due to the complex nature of the procedures and serious complications. In recent years, there has been increasing interest in the newer, less invasive superficial serratus block and combined serratus block. Serratus anterior plane block (SAPB) can be applied in two ways. Deep SPB (DSPB) is applied under the serratus anterior muscle, while superficial SPB (YSPB) is applied above the serratus anterior muscle. In recent years, deep + superficial SPB, or combined SPB (KSPB), has begun to be applied in order to increase the area of effect of local anesthetics and to prevent block failure. This study aims to compare superficial and combined serratus anterior plane blocks. Superficial serratus anterior plane block procedure: The USG probe is placed on the 4th rib in the mid-axillary line. After visualizing the muscle structures up to the rib (latissimus dorsi, teres major, and serratus anterior), the needle is advanced using the in-plane technique to the serratus anterior muscle, under the latissimus dorsi muscle, and hydrodissection is performed with 2 ml of saline to ensure positional accuracy. Then, 15 ml of 0.25% bupivacaine is injected into this area. KSAB procedure: The USG probe is placed on the 4th rib in the mid-axillary line. After visualizing the muscle structures up to the rib (latissimus dorsi, teres major, and serratus anterior), the needle is advanced using the in-plane technique to the 4th rib, under the serratus anterior muscle, and onto the rib. Hydrodissection is performed with 2 ml of saline to ensure positional accuracy. Then, 15 ml of 0.25% bupivacaine is injected into this area. The needle is then withdrawn 1-2 cm and positioned over the serratus anterior muscle, below the latissimus dorsi muscle. Hydrodissection with 2 ml of saline is performed to ensure accuracy. Then, 15 ml of 0.25% bupivacaine is injected into this area. A total of 30 ml of bupivacaine will be injected, and the procedure will be terminated. In our clinic, multimodal analgesia is preferred for patients undergoing mastectomy. Peripheral nerve blocks (for all suitable and consenting patients) are used in conjunction with intravenous analgesic agents. Both block types are routinely applied in suitable patients who have undergone mastectomy.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-80 years
* Individuals with ASA scores I-II-III
* Individuals with a Body Mass Index (BMI) between 18-40

Exclusion Criteria:

* Individuals under 18 years of age and over 80 years of age
* Individuals with an ASA score of IV or higher
* Individuals with advanced comorbidities
* Individuals with a history of bleeding diathesis
* Patients with infection in the area to be blocked
* Individuals with a BMI below 18 and above 40

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who undergone mastectomy surgery
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption | 24 hours postoperative
  Patients will be monitored for 24-hour opioid consumption with patient-controlled analgesia.

SECONDARY OUTCOMES:
Numeric Rating Scale (NRS) | 1 hour
  NRS is a scoring system ranging from 0 to 10, where higher values indicate a higher degree of pain.
  Pain level assessed by Numeric Rating Scale (NRS) in the first 24 hours postoperatively, pain at 1 hour, 2, 4, 12, and 24 hours, and pain with rest and coughing.
Numeric Rating Scale (NRS) | 2 hour
  NRS is a scoring system ranging from 0 to 10, where higher values indicate a higher degree of pain.
  Pain level assessed by Numeric Rating Scale (NRS) in the first 24 hours postoperatively, pain at 1 hour, 2, 4, 12, and 24 hours, and pain with rest and coughing.
Numeric Rating Scale (NRS) | 4 hour
  NRS is a scoring system ranging from 0 to 10, where higher values indicate a higher degree of pain.
  Pain level assessed by Numeric Rating Scale (NRS) in the first 24 hours postoperatively, pain at 1 hour, 2, 4, 12, and 24 hours, and pain with rest and coughing.
Numeric Rating Scale (NRS) | 12 hour
  NRS is a scoring system ranging from 0 to 10, where higher values indicate a higher degree of pain.
  Pain level assessed by Numeric Rating Scale (NRS) in the first 24 hours postoperatively, pain at 1 hour, 2, 4, 12, and 24 hours, and pain with rest and coughing.
Numeric Rating Scale (NRS) | 24 hour
  NRS is a scoring system ranging from 0 to 10, where higher values indicate a higher degree of pain.
  Pain level assessed by Numeric Rating Scale (NRS) in the first 24 hours postoperatively, pain at 1 hour, 2, 4, 12, and 24 hours, and pain with rest and coughing.
Patient satisfaction score | 24 hour
  Patient satisfaction will be evaluated using a 5-point Likert scale at 24 hours postoperatively.
  A Likert scale is a system of scores ranging from 1 to 5, where 1 (not satisfied at all) and 5 (very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Ozguner, Principal Investigator — Ankara Etlik City Hospital
Locations (1):
- Ankara Etlik City Hospital, Ankara, Varlık Mahallesi, Halil Sezai Erkut Caddesi Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chai B, Wang Q, Du J, Chen T, Qian Y, Zhu Z, Feng Z, Kang X. Research Progress on Serratus Anterior Plane Block in Breast Surgery: A Narrative Review. Pain Ther. 2023 Apr;12(2):323-337. doi: 10.1007/s40122-022-00456-z. Epub 2022 Dec 9. PMID 36484891
- [Result] Ozguner Y, Yazar CO, Aydin F, Zengin M, Arik E, Kotanoglu MS, Altinsoy S, Ergil J. Comparison of the analgesic efficacy of combined superficial and deep serratus anterior plane block versus pectoserratus plane block following modified radical mastectomy surgery. BMC Anesthesiol. 2025 Jul 28;25(1):358. doi: 10.1186/s12871-025-03213-9. PMID 40721998
- [Result] Ulger G, Zengin M, Kucuk O, Baldemir R, Kaybal O, Tunc M, Sazak H, Alagoz A. Comparison of combined deep and superficial serratus anterior block with thoracic paravertebral block for postoperative pain in patients undergoing video-assisted thoracoscopic surgery. Turk J Med Sci. 2024 Aug 4;54(5):1021-1032. doi: 10.55730/1300-0144.5881. eCollection 2024. PMID 39473759